CLINICAL TRIAL: NCT03142802
Title: Phase II Study of Effectiveness of Using Low-dose CT in Patient Undergoing Surveillance for Clinical Stage I Testicular Cancer
Brief Title: Low-Dose CT - Stage I Testicular Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 05-0436-CE
Record Dates: First submitted 2017-04-27; First posted 2017-05-05 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Testicular Cancer
Keywords: Testicular cancer; low-dose CT; CT scan
MeSH Terms: conditions — Testicular Neoplasms | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Intervention Model Description: Patients diagnosed with testicular germ cell cancer will undergo both standard and low dose CT scan of the abdomen and pelvis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with testicular germ cell cancer (Experimental): Patients with testicular germ cell cancer who have either been newly diagnosed, or have stage I cancer already on surveillance program will undergo conventional and low dose CT. Based on the imaging, they may undergo a surveillance program using low-dose CT.
  Interventions: Diagnostic Test: Low-dose computed tomography (LDCT)

INTERVENTIONS:
Diagnostic Test: Low-dose computed tomography (LDCT) — In phase A of the study, patients will undergo conventional CT along with low dose CT. If patients have a normal conventional CT and a satisfactory low dose CT, they will move onto Phase B of the study in which they will undergo surveillance using low-dose CT. Three outcomes are possible with low-dose CT surveillance:
  1. Normal LDCT:
     - Patient continues on the study (i.e. continued surveillance)
  2. Suspicious LDCT:
     - Will undergo conventional CT and if results are normal, patient will continue on study. If conventional CT is abnormal, they will be taken off study
  3. Elevated serum tumour markers or other evidence of metastatic disease:
     * Patient goes off study

SUMMARY:
Patients with primary germ cell cancer of the testicles confined to the testis can avoid adjuvant treatment by entering a surveillance protocol. In the surveillance protocol, patients are followed for up to ten years with serial computed tomography scans to detect recurrence. Multiple CT scans expose patients to a significant amount of radiation, which may be associated with an increased risk of secondary malignancies. This study hypothesizes that low dose CT scans are as effective as standard dose CT scans in detecting disease recurrence in this setting and will significantly reduce radiation exposure in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Phase A:
* Newly diagnosed testicular germ cell testicular cancer (GCT) with no clinical or tumour marker evidence of metastases
* Stage I disease according to UICC stage groupings and currently on surveillance (in Year 1 of non-seminoma surveillance or year 1 or 2 of seminoma surveillance)
* ECOG performance status 0 or 1
* Phase B:
* Stage I disease according to UICC stage Groupings
* Initial Low dose CT considered by study radiologist to be of sufficient quality to allow surveillance using LDCT protocol

Exclusion Criteria:

* any medical conditions that render the patient ineligible to undergo the protocol or procedure

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2005-09-16 (Actual); Primary Completion 2011-10-14 (Actual); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Difference in size of the retroperitoneal lymph node mass | 9 years
  The difference in size of lymph node mass at the time of relapse between low dose CT and conventional CT. This is to evaluate the effectiveness of using low-dose CT in patients undergoing surveillance.

SECONDARY OUTCOMES:
Time on surveillance | 6 years
  Amount of time patient is on surveillance before detection of relapse.
Amount of false positive rate of LDCTs | 6 years
Proportion of patients unsuitable for LDCT surveillance | 6 years
  Gather information on proportion of patients who were unsuitable for LDCT surveillance due to poor image quality
Proportion of patients who have to discontinue LDCT surveillance | 6 years
  Gather information on proportion of patients who had to discontinue LDCT surveillance due to poor image quality.
Amount of prospective identification of first modality to detect relapse | 6 years
  To prospectively identify the first modality to detect relapse (patient symptoms, clinical examination, tumour marker, imaging)
Proportion of disease-free survival | 6 years
  To document proportion of disease-free survival
Proportion of overall survival | 6 years
  To document proportion of overall survival
Amount of prospective documentation of treatment for testicular germ cell cancer relapse | 6 Years
  To prospectively document the treatment types for patients who have relapsed.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Chung, Principal Investigator — The Princess Margaret Cancer Foundation
Locations (1):
- University Health Network, Princess Margaret Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chung P, O'Malley ME, Jewett MAS, Bedard PL, Panzarella T, Sturgeon J, Moore MJ, Hamilton R, Hansen AR, Anson-Cartwright L, Gospodarowicz M, Warde P. Detection of Relapse by Low-dose Computed Tomography During Surveillance in Stage I Testicular Germ Cell Tumours. Eur Urol Oncol. 2019 Jul;2(4):437-442. doi: 10.1016/j.euo.2018.08.031. Epub 2018 Oct 2. PMID 31277780